CLINICAL TRIAL: NCT04631549
Title: A Multi-center, Non-randomized, Open-label, Parallel Controlled Pharmacokinetic Study of SHR3680 in Participants With Mild to Moderate Liver Impairment and Healthy Participants
Brief Title: An Investigational Study of SHR3680 in Participants With Mild to Moderate Liver Impairment and Healthy Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SHR3680-I-106
Record Dates: First submitted 2020-11-13; First posted 2020-11-17 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Hepatic Impairment; Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy participants (Experimental): Intervention: Drug: SHR3680 single dose
  Interventions: Drug: SHR3680
- Mild liver impairment (Experimental): Intervention: Drug: SHR3680 single dose
  Interventions: Drug: SHR3680
- Moderate liver impairment (Experimental): Intervention: Drug: SHR3680 single dose
  Interventions: Drug: SHR3680

INTERVENTIONS:
Drug: SHR3680 — SHR3680, PO, single dose

SUMMARY:
The purpose of this study is to investigate SHR3680 in participants with different levels of liver function

ELIGIBILITY:
Inclusion Criteria:

-

Participants with mild to moderate liver impairment must meet all of the following criteria to enter the study:

* The informed consent is signed before the trial, and the content, process and possible adverse reactions are fully understood; Be able to complete the study according to the requirements of the test scheme;
* Only for male, subjects aged 18 to 75 years (including both ends) on the date of signing informed consent;
* The body weight subjects is no less than 50 kg. Body mass index (BMI) is in the range of 19.0 kg/m2-29.0 kg/m2 (including the critical value);
* Primary liver disease (except for drug-induced liver injury) is necessary for patients with liver impairment, then patients with mild liver impairment (Child-Pugh score: 5-6) who are assessed as grade A according to Child-Pugh classification must be taken the clinical stability was ≥ 28 days before taking the experimental drug; while patients with moderate liver impairment (Child-Pugh score: 7-9) who are assessed as grade B according to Child-Pugh classification must be taken the clinical stability was ≥ 14 days before taking the experimental drug;
* Patients who have stable medication regimen for liver impairment, complications and other concomitant diseases within at least 28 days before taking the experimental drug, and the medication does not need to be adjusted (including drug type, dosage or frequency) during the clinical trials; or those who do not use the drug;
* The function of vital organs meets the following criteria: Absolute neutrophil count (ANC) ≥ 1.0 × 109 / L (1000 / mm3); Hemoglobin (Hgb) ≥ 9.0 g / dL (90g / L); Platelet ≥ 75.0 × 109 / L (75000 / mm3); Creatinine clearance rate (CLcr) ≥ 80 mL / min; The corrected QTc interval (QTcF) was less than 450 msec (male);
* In addition to liver impairment and complications, the investigator judged good condition according to the history inquiry, vital signs, physical examination, routine laboratory examination, 12-lead ECG, abdominal ultrasound scan, EEG, etc., and there was no other clinically significant abnormality;
* Male subjects are willing to have no family planning during the trial and within 6 months after the last administration of the trial drug, and voluntarily take effective contraceptive measures, or have undergone surgical sterilization.

Exclusion Criteria:

-

Participants with mild to moderate liver impairment who meet any of the following criteria will not be eligible for this study:

* Subjects had any of the following conditions: Patients with hepatic encephalopathy (according to Child-Pugh score); previous liver transplantation; severe portal hypertension or portal systemic shunt; suspected or diagnosed liver cancer or other malignant tumors; liver failure patients; esophageal and gastric variceal bleeding; severe / advanced ascites; hepatorenal syndrome patients; biliary tract Liver cirrhosis, biliary obstruction, cholestatic liver disease and other diseases that seriously affect bile excretion;
* In addition to the diseases leading to the diagnosis of liver impairment, the patients with severe acute and chronic diseases of other important organs within one year before screening, including but not limited to neuropsychiatric, digestive tract, respiratory system, urinary, endocrine, blood, immune and other diseases, were judged by the researchers to be unsuitable for the trial;
* Any of the following conditions occurred within 6 months prior to the study: myocardial infarction, congenital long QT syndrome, torsade de pointes (including persistent ventricular tachycardia and ventricular fibrillation), right bundle branch block and left anterior half block (bifascilar block), unstable angina pectoris, coronary / peripheral artery bypass grafting, and congestive heart failure syndrome (Grade III or IV according to NYHA), cerebrovascular accident, transient ischemic attack, or pulmonary embolism;
* Patients who had serious gastrointestinal diseases (except secondary gastrointestinal diseases caused by hepatitis) or had digestive system surgery 3 months before screening, and the researchers considered that drug absorption was affected;
* Warfarin or related coumarins were used for anticoagulant therapy within one month before screening, or warfarin or related coumarins were required for anticoagulant therapy during the trial period;
* During the screening period, liver function fluctuations (such as active hepatitis), rapid deterioration (such as advanced ascites, fever, active gastrointestinal bleeding), NCI CTCAE grade 2 or above, ongoing arrhythmia, and atrial fibrillation of any level occurred;
* People with allergic constitution, including those with severe drug allergy or history of drug allergy, and patients known to be allergic to the study drug SHR3680 or any excipients of the product;
* Those who have a history of drug use, or have a history of drug abuse in the past five years, or have a positive drug screening (except those with drug screening positive due to concomitant drug use);
* HIVAb positive, syphilisAb positive;
* Patients who have taken any clinical trial drugs within 3 months before screening; 14) Patients who had received drugs with definite potential hepatotoxicity and used them continuously for 7 days or more within 3 months before taking experimental drug;
* In 2 weeks before screening, they used traditional Chinese medicine (Chinese herbal medicine, Chinese patent medicine), dietary supplements and vitamins;
* Subjects with other factors not suitable to participate in this study were considered by the investigator.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Cmax | Day1~Day29
  Maximum concentration
AUC0-t | Day1~Day29
  Area under the concentration time curve from time zero to time t
AUC0-∞ | Day1~Day29
  Area under the concentration time curve extrapolated to infinity

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Eighth People'S Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No